CLINICAL TRIAL: NCT02057783
Title: Comparison of Standard Treatment by Continuous Positive Airway Pressure (CPAP) and CPAP Combined to a Physical Activity Program for Reducing Blood Pressure in Sleep Apnea Patients With Resistant Hypertension: RAP Randomized Controlled Trial
Brief Title: Physical Activity Program for Reducing Blood Pressure in Sleep Apnea Patients With Resistant Hypertension
Acronym: RAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AGIR à Dom (Other)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-AGIR-04
Record Dates: First submitted 2014-02-04; First posted 2014-02-07 (Estimated); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Hypertension, Resistant to Conventional Therapy; Sleep Apnea
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; Sleep Apnea Syndromes | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Physical activity (Experimental): Obstructive sleep apnea and resistant hypertension controlled + physical activity
  Interventions: Other: Physical activity
- Control Group (No Intervention): Obstructive sleep apnea and resistant hypertension controlled

INTERVENTIONS:
Other: Physical activity — Physical activity will carry out 3 times per week during 12 weeks for intervention arm
  Arms: Physical activity

SUMMARY:
Investigators hypothesize that CPAP treatment for suppressing OSAS in combination with a physical activity program will optimize 24-hour blood pressure control in patients with OSA-related resistant hypertension.

DETAILED DESCRIPTION:
1. Sleep apnea syndrome, resistant hypertension and cardio-vascular risk. There are many epidemiological and clinical cohort studies demonstrating an increasing cardiovascular risk associated with Obstructive Sleep Apnea Syndrome (OSAS). In epidemiological studies, OSA severity and incident hypertension are linked in a dose-response fashion. This is true even when taking into account usual confounding factors such as age, alcohol, tobacco consumption and body mass index. More specifically, OSAS is the leading cause of refractory hypertension and OSAS prevalence is up to 80% in patients with resistant hypertension.
2. CPAP treatment impact for reducing blood pressure in OSAS patients with resistant hypertension A recent small sample size randomized trial (n=35) demonstrated the positive impact of CPAP in decreasing both clinical and 24-hour ambulatory blood pressure. Compared to the control group, awake systolic/diastolic ambulatory blood pressure monitoring decreased significantly in the continuous positive airway pressure group (Delta: +3.1±3.3 /+2.1±2.7 vs. -6.5±3.3/ 4.5±1.9mmHg in control and CPAP groups respectively, p<0.05). Interestingly, the blood pressure changes were only observed while patients were awake, but not during nocturnal ambulatory blood pressure monitoring (Delta: +2.8±4.5/+1.8±3.5 vs. +1.6±3.5/+0.8±2.9mmHg, p=NS).

   HIPARCO Study, the largest Randomized Clinical Trial (RCT) in the field (n=194) recently published in JAMA (9 December 2013) also showed a significant but limited impact of CPAP on blood pressure. In an Intention To Treat analysis, CPAP significantly improved 24-h mean BP (3.0 mmHg; 95% CI 0.3 to 5.8; p=0.031) and DBP (3.2 mmHg; 95% CI 1.0 to 5.4; p=0.005) but not SBP (3.1; 95% CI -0.6 to 6.7; p=0.098). Moreover, patients in the CPAP group had 2.4 (1.2-5.1; p=0.019) times greater probability of recovering their dipper pattern. As CPAP alone is not enough in OSAS to sufficiently improve BP, further studies should address the efficacy of combined therapies in OSAS patients with resistant hypertension.
3. Resistant hypertension and physical activity A study has recently explored the impact of a standardized exercise program in patients suffering from resistant hypertension7. In this RCT, the authors have demonstrated that the group of patients who have benefit from a physical activity program had their systolic and diastolic 24-hour ambulatory blood pressure monitoring decreasing by 6±12 and 3±7 mmHg respectively(p=0.03). Thus, the physical activity implemented in this population enabled a better control of blood pressure values. However the authors do not give any information about the presence of the absence of Sleep Apnea Syndrome (SAS) in this cohort.
4. Study hypothesis:

Investigators hypothesize that CPAP treatment for suppressing OSAS in combination with a physical activity program will optimize 24-hour blood pressure control in patients with OSA-related resistant hypertension.

Originality: Up to now no study has assessed the effects of combining physical activity with CPAP treatment in patients with sleep apnea and resistant hypertension. Our work is will be the first aiming at evaluating the benefit of this combination on the control of the systolic blood arterial pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an obstructive sleep apnea (apnea-hypopnea index > or equal to 15)
* Patient with resistant hypertension uncontrolled by 3 or more antihypertensive agents
* Ambulatory patient

Exclusion Criteria:

* Acute hepatic failure, biliary cirrhosis, cholestasis
* Acute hypertension (SBP>= 180 mmHg and/or DBP >= 110 mmHg)
* Contraindication to CPAP treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-03-26 (Actual); Primary Completion 2025-02-18 (Estimated); Study Completion 2025-02-18 (Estimated)

PRIMARY OUTCOMES:
Systolic arterial blood pressure assessed by 24-hours home blood pressure monitoring | To baseline at 12 weeks
  Systolic arterial blood pressure assessed by 24-hours home blood pressure monitoring

SECONDARY OUTCOMES:
diastolic arterial blood pressure assessed by 24-hours home blood pressure monitoring | To baseline at 12 weeks
  diastolic arterial blood pressure assessed by 24-hours home blood pressure monitoring
Mean arterial blood pressure assessed by 24-hours home blood pressure monitoring | To baseline at 12 weeks
  Mean arterial blood pressure assessed by 24-hours home blood pressure monitoring
Change in physical activity: number of hour per day of physical activity | To baseline at 12 weeks
  Change in physical activity: number of hour per day of physical activity
pulse wave velocity | To baseline at 12 weeks
  pulse wave velocity
Change in physical activity : Metabolic Equivalents (METS) | To baseline at 12 weeks
  Change in physical activity : Metabolic Equivalents (METS)
Change in physical activity : Number of steps per day | To baseline at 12 weeks
  Change in physical activity : Number of steps per day
Change in sleep duration: Sleep to lying position duration ratio | To baseline at 12 weeks
  Change in sleep duration: Sleep to lying position duration ratio

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pépin, Pr MD PhD, Principal Investigator — Laboratoire EFCR, CHU de Grenoble, 38043, Grenoble, France
Locations (5):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec, Canada
- France (2):
  - Hopital Universitaire de Grenoble, La Tronche
  - Clinique Pasteur, Toulouse
- Switzerland (2):
  - Hopitaux Universitaires de Genève, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne